CLINICAL TRIAL: NCT02485392
Title: A Comparison of Robot-assisted Single Site and Laparoscopic Single-incision Cholecystectomy for Benign Gallbladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEK-ZH 2014-0114
Record Dates: First submitted 2015-02-19; First posted 2015-06-30 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Benign Gallbladder Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-Site robot-assisted cholecystectomy (Active Comparator): Single-Site robot-assisted cholecystectomy
  Interventions: Device: Da Vinci Single Site Robot-Assisted Cholecystectomy
- Single-incision laparoscopic cholecystectomy (Active Comparator): Single-incision laparoscopic cholecystectomy
  Interventions: Device: Single Incision Laparoscopic Cholecystectomy

INTERVENTIONS:
Device: Da Vinci Single Site Robot-Assisted Cholecystectomy
  Arms: Single-Site robot-assisted cholecystectomy
Device: Single Incision Laparoscopic Cholecystectomy
  Arms: Single-incision laparoscopic cholecystectomy

SUMMARY:
A single-blinded randomized clinical trial (RCT) designed to compare Single-Site robot-assisted with single-incision laparoscopic cholecystectomy. The study directly compares both surgical approaches in a cohort of 60 patients (30 patients in each arm) with benign gallbladder disease from the Department of Surgery at the Cantonal Hospital of Winterthur (Kantonsspital Winterthur) in Switzerland. The primary endpoint of the study is the surgeon's physical and mental stress load at the time of surgery and is assessed by validated Local Experienced Discomfort (LED) and Subjective Mental Effort Questionnaire (SMEQ) visual analogue scales. The secondary endpoints include costs of the procedure, intra-operative blood loss, operating time, intra-operative conversion rate and additional trocar placement, complications, length of hospital stay, Health-Related Quality of Life (HRQoL) and cosmesis. HRQoL and cosmesis will be assessed using the validated Gastrointestinal Quality of Life Index (GIQLI) and the Body Image Questionnaires (BIQ), respectively. The inclusion criteria cover most notably symptomatic cholecystolithiasis, chronic cholecystitis, benign gallbladder polyps and age ≥18 years. The exclusion criteria are, among others, acute cholecystitis, emergency cholecystectomy, previous extensive upper abdominal surgery and suspicion of malignant disease. Non-stratified block randomization (random block sizes 2 and 4) will be used to achieve balance in the allocation of participants to both treatments arms and prevent a premature decoding of the randomization scheme. Hereby, the patient will not be informed about the group assignment until the last outpatient follow-up and only after he/she has completed and returned all required questionnaires (GIQLI and BIQ). The operation will be performed according to the group assignment by senior surgeons only who have a wide experience in both robotic Single-Site and conventional single-incision laparoscopy. All data are recorded safely using the SecuTrialTM program. Sample-size calculations are based on the results of the previously mentioned experimental setup by Schatte et al, utilizing an estimated effect size of 0.8, at a power of 0.8 and an alpha-error level of 0.05, as well as considering a potential additional error margin of 10-15% of the calculations (G-Power 3.1 software, Heinrich-Heine University Duesseldorf/Germany). The estimated total duration of the study is 1.5 years, including the scheduled 1-month and 1-year postoperative follow-up visits. The study will be carried out in accordance with principles enunciated in the current version of the Declaration of Helsinki, the guidelines of Good Clinical Practice (GCP) issued by International Conference on Harmonization (ICH), and Swiss regulatory authority's requirements.

ELIGIBILITY:
Inclusion Criteria:

* Patient compliance and geographic proximity allow proper preoperative checkup and postoperative follow-up
* Written informed consent given by the patient
* Women who are not breastfeeding and are not pregnant
* Age ≥18 years
* Symptomatic cholecystolithiasis
* Chronic cholecystitis
* Benign gallbladder polyps

Exclusion Criteria:

* Significant concomitant diseases making the patient unsuitable for abdominal surgery by the judgement of the physicians involved
* Peritoneal carcinomatosis or other extensive metastatic disease
* American Society of Anesthesiologists (ASA) IV and V patients
* Mental or organic disorders which could interfere with giving informed consent or receiving treatments
* Contraindications to pneumoperitoneum
* Suspicion of malignant disease
* Previous extensive upper abdominal surgery
* Acute cholecystitis
* Emergency cholecystectomy
* Obesity II°---III° (BMI>35.0 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Surgeon's comfort as measured by LED and SMEQ questionnaires | 1 Day

SECONDARY OUTCOMES:
Intra-operative blood loss | 1 day
Operating time | 1 day
Intra--operative conversion rate | 1 day
Complications | 1 year
Length of hospital stay | until discharge (average of 2 days)
Costs of procedure | until discharge (average of 2 days)
Health--Related Quality of Life (HRQoL) | 1 year
Cosmesis as measured by Body Image Questionnaire (BIQ) | 1 year
Intra-operative additional trocar placement | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Breitenstein, MD, Principal Investigator — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital Winterthur, Winterthur, Switzerland

REFERENCES:
- [Derived] Grochola LF, Soll C, Zehnder A, Wyss R, Herzog P, Breitenstein S. Robot-assisted versus laparoscopic single-incision cholecystectomy: results of a randomized controlled trial. Surg Endosc. 2019 May;33(5):1482-1490. doi: 10.1007/s00464-018-6430-7. Epub 2018 Sep 14. PMID 30218263
- [Derived] Grochola LF, Soll C, Zehnder A, Wyss R, Herzog P, Breitenstein S. Robot-assisted single-site compared with laparoscopic single-incision cholecystectomy for benign gallbladder disease: protocol for a randomized controlled trial. BMC Surg. 2017 Feb 9;17(1):13. doi: 10.1186/s12893-017-0206-1. PMID 28183345